CLINICAL TRIAL: NCT07321652
Title: Phase III Evaluation of Fixed Duration Zanubrutinib Plus Sonrotoclax-Based Therapy Compared to Continuous Zanubrutinib in Previously Untreated Older Patients With Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma (CLL/SLL)
Brief Title: Testing the Addition of Anti-Cancer Drug Sonrotoclax, to the Standard Treatment Zanubrutinib, for Previously Untreated CLL/SLL
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A042302
Record Dates: First submitted 2026-01-05; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Chronic Lymphocytic Leukemia; Small Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — zanubrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1 (zanubrutinib) (Active Comparator): Patients receive zanubrutinib PO BID on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo restaging starting at cycle 15 day 1. Patients with at least partial remission continue therapy as described above. Patients with progressive disease proceed to follow up. Patients undergo CT scan, bone marrow aspiration and blood sample collection throughout the study.
  Interventions: Drug: Zanubrutinib; Procedure: Computed Tomography; Procedure: Bone Marrow Aspiration; Procedure: Biospecimen Collection; Other: Survey Administration
- Arm 2 (zanubrutinib and sonrotoclax) (Experimental): Patients receive zanubrutinib PO BID on days 1-28 of each cycle. Starting cycle 4 day 1 patients also receive sonrotoclax PO QD on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo restaging starting at cycle 15 day 1. Patients with undetectable MRD and a response of PR, PR-L, CR, CCR or CRi stop therapy at cycle 15 day 28 and proceed to follow up. Patients with detectable MRD and an objective response to therapy are re-randomized to arm 2B or arm 2C.
  ARM 2B: Patients continue zanubrutinib PO BID sonrotoclax PO QD on days 1-28 of each cycle. Cycles repeat every 28 days for an additonal 12 cycles in the absence of disease progression or unacceptable toxicity.
  ARM 2C: Patients discontinue therapy starting at cycle 15 day 28 and proceed to follow up.
  Patients undergo CT scan, bone marrow aspiration and blood sample collection
  Interventions: Drug: Zanubrutinib; Drug: Sonrotoclax; Procedure: Computed Tomography; Procedure: Bone Marrow Aspiration; Procedure: Biospecimen Collection; Other: Survey Administration

INTERVENTIONS:
Drug: Zanubrutinib — Given PO
Drug: Sonrotoclax — Given PO
  Arms: Arm 2 (zanubrutinib and sonrotoclax)
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CT Scan; Cat Scan
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspiration
Procedure: Biospecimen Collection — Undergo blood sample collection
Other: Survey Administration — Ancillary studies

SUMMARY:
This phase III trial compares the effect of adding sonrotoclax to zanubrutinib versus zanubrutinib alone for the treatment of patients with untreated chronic lymphoblastic leukemia (CLL)/small lymphocytic lymphoma (SLL). Sonrotoclax is in a class of medications called B-cell lymphoma-2 (BCL-2) inhibitors. It may stop the growth of cancer cells by blocking Bcl-2, a protein needed for cancer cell survival. Zanubrutinib is in a class of medications called kinase inhibitors. It blocks a protein called BTK, which is present on B-cell (a type of white blood cells) cancers such as mantel cell lymphoma at abnormal levels. This may help keep cancer cells from growing and spreading. Giving sonrotoclax and zanubrutinib may be more effective than zanubrutinib alone for the treatment of untreated CLL/SLL.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare the progression free survival (PFS) between minimal residual disease (MRD)-guided zanubrutinib sonrotoclax therapy to continuous zanubrutinib as control.

II. To determine the PFS comparing fixed duration zanubrutinib sonrotoclax therapy to continuous zanubrutinib as control.

SECONDARY OBJECTIVES:

I. To compare the PFS between the patients with MRD-detectable disease treated with fixed duration zanubrutinib sonrotoclax to the PFS of the patients with MRD detectable disease who receive one additional year of combination therapy.

II. To determine the overall survival of all arms of the study. III. To determine the frequency of patients with MRD-detectable disease who convert to undetectable MRD, and at what depth and for how long, after receiving an extra year of combination therapy on the MRD-guided zanubrutinib sonrotoclax therapy arm.

IV. To determine and compare the overall response rate (ORR defined as PR, CR, CCR, CRi) and complete remission rate (CR) after 14 cycles of therapy among the three arms.

V. To compare time to the next CLL/SLL therapy among treatment arms. VI. To determine the rates and severity of toxicity in each arm, with a particular focus on adverse events of special interest that include infections, cardiovascular events (arrhythmias, heart failure, hypertension), tumor lysis syndrome, bleeding events, cytopenias, and second malignancies.

VII. To compare patient-reported symptomatic adverse events as assessed by the Patient Reported Outcome-Common Terminology Criteria for Adverse Events (PRO-CTCAE) between arms 1 and 2.

EXPLORATORY OBJECTIVES:

I. To compare the best achieved rate of undetectable MRD (uMRD) between the fixed duration zanubrutinib sonrotoclax arm and the MRD guided zanubrutinib sonrotoclax arm.

II. To compare rates of undetectable MRD measured by the immunoglobulin heavy chain (IGH) sequencing assay ClonoSeq (sensitivity 1 in 10^-6) to undetectable MRD measured by standard six-color flow cytometry (uMRD4), and to compare results from bone marrow to peripheral blood.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM 1: Patients receive zanubrutinib orally (PO) twice daily (BID) on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo restaging starting at cycle 15 day 1. Patients with at least partial remission continue therapy as described above. Patients with progressive disease proceed to follow up. Patients undergo computed tomography (CT) scan, bone marrow aspiration and blood sample collection throughout the study.

ARM 2: Patients receive zanubrutinib PO BID on days 1-28 of each cycle. Starting cycle 4 day 1 patients also receive sonrotoclax PO daily (QD) on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo restaging starting at cycle 15 day 1. Patients with undetectable MRD and a response of PR, partial response with persistent lymphocytosis (PR-L), CR, CCR or CRi stop therapy at cycle 15 day 28 and proceed to follow up. Patients with detectable MRD and an objective response to therapy are re-randomized to arm 2B or arm 2C.

ARM 2B: Patients continue zanubrutinib PO BID sonrotoclax PO QD on days 1-28 of each cycle. Cycles repeat every 28 days for an additonal 12 cycles in the absence of disease progression or unacceptable toxicity.

ARM 2C: Patients discontinue therapy starting at cycle 15 day 28 and proceed to follow up.

Patients undergo CT scan, bone marrow aspiration and blood sample collection throughout the study.

After completion of study treatment, patients are followed up every 3 months for 3 years then every 6 months until 10 years for study registration. Patients with progression or the start of non protocol CLL directed therapy are followed every 6 months for 10 years from registration.

ELIGIBILITY:
Inclusion Criteria:

* STEP 0: This bone marrow or peripheral blood submission to Adaptive is mandatory prior to registration/randomization for real-time identification of the clone needed for MRD testing. The bone marrow sample should be from the first aspiration (i.e., first pull). Aspirate needle should be redirected if needed to get first pull bone marrow aspirate. It should be obtained as soon after pre-registration as possible to confirm registration eligibility
* STEP 0: Patients must be diagnosed with CLL/SLL according to International Workshop on Chronic Lymphocytic Leukemia (IWCLL) 2018 criteria that includes all of the following:

  * ≥ 5 x10^9 /L B lymphocytes (5000/μL) in the peripheral blood (CLL) or a lymph node biopsy demonstrating SLL with the below immunophenotype (SLL)
  * On morphologic review, the leukemic cells must be small mature lymphocytes
  * Immunophenotype of CLL cells (performed locally) must reveal a clonal B-cell population, which coexpress the B cell surface markers of CD19 and CD20, as well as the T-cell antigen CD5. Patients with bright surface immunoglobulin expression or lack of CD23 expression in > 10% of cells must lack t(11;14) translocation by interphase cytogenetics
* STEP 0: Patients must meet criteria for treatment as defined by IWCLL 2018 guidelines which includes at least one of the following criteria:

  * Evidence of marrow failure as manifested by the development or worsening of anemia or thrombocytopenia (not attributable to autoimmune hemolytic anemia or thrombocytopenia), typically hemoglobin (Hb) < 10 g/dL, platelet count < 100,000/mm^3
  * Massive (> 6 cm below the costal margin), progressive or symptomatic splenomegaly
  * Massive nodes (ie, > 10 cm in longest diameter) or progressive or symptomatic lymphadenopathy
  * Autoimmune anemia and/or thrombocytopenia that is poorly responsive to standard therapy
  * Constitutional symptoms, which include any of the following:

    * Unintentional weight loss of ≥ 10% within the previous 6 months
    * Significant fatigue (ie. Eastern Cooperative Oncology Group [ECOG] performance status [PS] ≥ 2)
    * Fevers >100.5 °F or 38.0°C for 2 weeks or more without evidence of infection
    * Night sweats > 1 month without evidence of infection
* STEP 0: Patients must not have had prior therapy for CLL (except palliative steroids or treatment of autoimmune complications of CLL with rituximab or steroids)
* STEP 0: Treatment with rituximab and/or high-dose corticosteroids for autoimmune complications of CLL must be completed prior to enrollment. Palliative steroids must be at a dose not higher than 20 mg/day of prednisone or equivalent corticosteroid at the time of registration
* STEP 0: Age ≥ 65 years
* STEP 0: ECOG performance status ≤ 2
* STEP 0: Patients with known HIV infection on effective anti-retroviral therapy with undetectable viral load within 6 months prior to registration are eligible for this trial
* STEP 0: For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* STEP 0: Patients with a history of hepatitis C virus (HCV), infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* STEP 0: Patients must not be receiving active systemic anticoagulation with warfarin. Patients must be off warfarin therapy for at least 5 half-lives washout and with normal INR prior to enrollment
* STEP 0: Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients must be class 2B or better.

Patients with acute cardiac events within 6 months prior to registration should be carefully evaluated for their suitability for enrollment

* STEP 0: No patients with a history of a severe bleeding disorder or a history of hemorrhagic stroke or intracranial hemorrhage
* STEP 0: No patients with known active progressive central nervous system (CNS) disease
* STEP 0: No known medical condition causing an inability to swallow oral formulations of agents
* STEP 1: The adaptive report confirming a measurable and trackable B cell clone
* STEP 1: Patients may not have had major surgery within 7 days of enrollment, or minor surgery within 5 days of enrollment. Examples of minor surgery include dental surgery, insertion of a venous access device, skin biopsy, or aspiration of a joint. The decision about whether a surgery is major or minor can be made at the discretion of the treating physician
* STEP 1: No patients with ongoing active fungal, bacterial or viral infection requiring systemic therapy except those described in the protocol document
* STEP 1: Patients must not require more than 20 mg prednisone or equivalent corticosteroid daily
* STEP 1: Patients must not have uncontrolled active systemic infection requiring intravenous antibiotics
* STEP 1: Patients must not have continued requirement for therapy with a strong CYP3A4/5 inhibitor or inducer. Any such inhibitor or inducer must have been discontinued at least 14 days or 5 half-lives (whichever is shorter) before the first dose of study drug
* STEP 1: Absolute neutrophil count (ANC) ≥ 1,000/mm3 unless due to marrow involvement
* STEP 1: Platelet count ≥ 30,000/mm3
* STEP 1: Total bilirubin ≤ 1.5 x upper limit of normal (ULN) (unless due to liver involvement, hemolysis or Gilbert's disease)
* STEP 1: Aspartate aminotransferase (AST)(serum glutamic oxaloacetic transaminase [SGOT])/ alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) ≤ 3.0 x upper limit of normal (ULN) unless due to disease infiltration of the liver
* STEP 1: Calculated (calc.) creatinine clearance by Chronic Kidney Disease Epidemiology Collaboration equation (CKD-EPI) ≥ 30 mL/min
* STEP 1: Urine protein to creatinine ratio < 1 or urine protein ≤ 1+
* STEP 2: Detectable MRD ≥ 10 residual clonal cells per million nucleated cells in peripheral blood at the C15 restaging evaluation from ClonoSEQ
* STEP 2: Response of PR, PR-L, CR, CCR or CRi to zanubrutinib sonrotoclax therapy

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 466 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2028-09-30 (Estimated); Study Completion 2038-09-30 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | From initial randomization date until the earlier of disease progression or death from any cause, up to 10 years
  From initial randomization date until the earlier of disease progression or death from any cause. PFS estimates for zanubrutinib plus sonrotoclax therapy to continuous Zanubrutinib.

OTHER OUTCOMES:
PFS for patients with MRD detectable disease treated with fixed duration zanubrutinib sonrotoclax versus patients with MRD detectable disease who receive one additional year of combination therapy | up to 10 years
  Undetectable (u) MRD will be defined as < 10 in 1,000,000 (less than 1 in 10^-5 [uMRD5]) on peripheral blood, and the depth of response below that level, (i.e. down to 10^-6 [uMRD6]), will also be collected. Kaplan-Meier will be used to estimate survival curves, log-rank tests to compare between survival curves, and hazard ration (HRs) and associated 95% CIs will be reported.
Overall survival | Up to 10 years
  OS will be summarized using Kaplan-Meier methodology, with hazard ratios from a stratified Cox proportional hazards model and log-rank test results provided.
Percentage of patients with MRD detectable disease who convert to uMRD after receiving an extra year of combination therapy on the MRD-guided Zanubrutinib sonrotoclax therapy arm | Up to 10 years
  Proportions of number of MRD+ to uMRD conversion by total number of evaluable patients will be estimated with their corresponding 95% CIs.
Overall response rate among treatment arms | Up to 10 years
  Overall response rate is defined as the highest response achieved during the first 15 cycles of treatment. A response is defined as a patients achieving PR+.
Time to next CLL/SLL therapy | Up to 10 years
  Kaplan-Meier estimates and 95% CIs of TTNT. Time is measured as the time from the end of initial treatment to the initiation of subsequent treatment.
Adverse Event Rates and Severity | Up to 10 years
  Frequency and severity of adverse events and tolerability for each embedded treatment regimen will be collected and summarized using descriptive statistics.
Patient-reported symptomatic adverse events | Up to 10 years
  As assessed by the Patient Reported Outcome-Common Terminology Criteria for Adverse Events, the frequency and proportion of patients with a maximum baseline-adjusted composite score greater than 0 will be compared between arms using Fisher's exact test. Similarly, the frequency and proportion of patients with a maximum baseline-adjusted composite score greater than or equal to 3 will be compared between arms using Fisher's exact test.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer R Brown, MD, Study Chair — Alliance for Clinical Trials in Oncology

IPD SHARING:
Plan to Share IPD: No